CLINICAL TRIAL: NCT01301820
Title: Phase II Multicentric Trial Maintenance Therapy With 6 Monthly Revlimid® Cycles Alternated With 6 Monthly Vidaza® Cycles in First CR After Induction LIA Chemotherapy for Elderly Fit Patients With Poor Prognosis Acute Myeloid Leukemia.
Brief Title: Elderly Patients With Acute Myeloid Leukemia (AML), Maintenance Phase After Complete Remission (CR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAMSA-maintenance Rev-5Aza
Record Dates: First submitted 2011-02-04; First posted 2011-02-23 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: maintenance treatment; Disease free survival
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Other): maintenance study treatment: azacitidine sc 75 mg/m²/d (d1- d7) in first cycle: months 1,3,5,7,9 ,11 then lenalidomide 10mg/d (d1- d21) months 2,4,6,8,10,12
  Interventions: Drug: azacitidine
- ARM B (Other): maintenance study treatment: lenalidomide 10mg/d (d1- d21)in first cycle and months 1,3,5,7,9 ,11 then azacitidine sc 75 mg/m²/d (d1- d7) months 2,4,6,8,10,12
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: azacitidine — azacitidine sc 75 mg/m²/d (d1- d7)
  Other Names: vidaza®
  Arms: ARM A
Drug: Lenalidomide — lenalidomide 10mg/d (d1- d21)
  Other Names: revlimid®
  Arms: ARM B

SUMMARY:
Phase II Multicentric Trial Open Label, Multicenter, randomized to evaluate the efficacy of a Maintenance Therapy in First Complete Remission After Induction for Elderly (≥ 60) Fit Patients With Poor Prognosis Acute Myeloid Leukemia (AML).

The disease-free survival (DFS) of the patients included in this study will be compared to the ones of the two previously reported groups of patients treated with the same LIA induction therapy

DETAILED DESCRIPTION:
* The primary objective of this study will be to improve the DFS with an alternate schema combining azacitidine and lenalidomide in elderly fit patients with previously untreated AML and with high risk cytogenetics or secondary AML, who achieved either a complete remission after an LIA induction therapy
* The secondary objectives will be to determine the relapse incidence, overall survival, event free survival at 1 and 2 years of follow-up, toxicities of the treatment, incidence of infectious events.
* To define a gene expression and promoter methylation signatures associated with CR and absence of relapse when patients received azacitidine and lenalidomide. Gene promoter methylation and gene expression profiling will be performed at diagnosis, at CR, and after 2 courses of azacitidine and lenalidomide in order to give insight within the mechanisms involved by the use of these 2 drugs and to identify new epigenetic prognostic markers.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed acute myeloid leukemia (AML) with :

  * At least 60 years of age and fit for intensive chemotherapy: PS <2 (ECOG)
  * Absence of significant co-morbidities
  * Less than 75 years* of age
  * LAM with high risk features (blasts > 20% in bone marrow)
  * Poor risk cytogenetics
  * Life expectancy > 1 month
  * Affiliated to social security regimen
  * No granulocytic sarcoma as sole site of disease
  * Able and willing to provide written and signed informed consent

Exclusion Criteria:

* Total bilirubin > 2 times upper limit of normal
* AST and ALT and/or alkaline phosphatase > 4 times upper limit of normal if not in relation with AML.
* Factor V < 50% without DIC (Disseminated Intravascular Coagulation)
* NYHA class III or IV congestive heart failure (Echo < 40%, LVEF < 50%),Unstable angina pectoris, Serious cardiac arrhythmia
* Renal failure not related to AML: serum creatinin > 170 μmol/L or clearance of creatinin ≤ 50 mL/mn
* Known HIV 1- HIV 2 positivity
* Prior therapy with azacitidine or lenalidomide
* Psychiatric illness or social situations that would preclude compliance with study requirements
* Uncontrolled infection
* Urgent chemotherapy for DIC, spontaneous tumoral lyse syndrome, leucostase without cytogentic results
* Women who are pregnant or breastfeeding
* Women who are unwilling or unable to use an acceptable contraceptive method to avoid pregnancy
* Men who are unwilling or unable to use an acceptable method of birth control

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
DFS | 18 months
  The primary objective of this study will be to improve the DFS with an alternate schema combining azacitidine and lenalidomide in elderly fit patients with previously untreated AML and with high risk cytogenetics or secondary AML, who achieved either a complete remission after an LIA induction therapy.

SECONDARY OUTCOMES:
relapse incidence OS EFS Infectious events | until death
  The secondary objectives will be to determine the relapse incidence, overall survival, event free survival at 1 and 2 years of follow-up, toxicities of the treatment, incidence of infectious events.
gene expression and promoter methylation signatures associated with CR | 0
  To define a gene expression and promoter methylation signatures associated with CR and absence of relapse when patients received azacitidine and lenalidomide. Gene promoter methylation and gene expression profiling will be performed at diagnosis, at CR, and after 2 courses of azacitidine and lenalidomide in order to give insight within the mechanisms involved by the use of these 2 drugs and to identify new epigenetic prognostic markers.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde HUNAULT BERGER, MD PD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Mathilde HUNAULT BERGER, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FILO Website — http://www.filo-leucemie.org